CLINICAL TRIAL: NCT07360730
Title: Prospective Multicentre Registry of High-Purity Type I Collagen Nerve Wrapping in Peripheral Nerve Procedures: Early Clinical Outcomes
Brief Title: High-Purity Type I Collagen Nerve Wrapping in Peripheral Nerve Procedures: A Prospective Registry
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adichunchanagiri Institute of Medical Sciences, B G Nagara (Other)
Collaborators: Mysore Medical College and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIMS/IEC/269/2025
Record Dates: First submitted 2026-01-02; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Nerve Injuries; Neuroma of Nerve Repair; Nerve Graft; Complications, Mechanical; Peripheral Nerve Decompression Injury; Neuroma
MeSH Terms: conditions — Peripheral Nerve Injuries; Neuroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPTC Nerve Wrap Arm (Experimental): Participants undergoing peripheral nerve procedures-including nerve repair, coaptation, grafting, nerve transfer, or decompression-in whom a High-Purity Type I Collagen (HPTC) membrane is used intraoperatively as a circumferential nerve wrap. Outcomes related to motor recovery, sensory recovery, neuropathic pain, complications, and patient-reported functional status are prospectively assessed.
  Interventions: Device: High-Purity Type I Collagen (HPTC) Nerve Wrap

INTERVENTIONS:
Device: High-Purity Type I Collagen (HPTC) Nerve Wrap — After completion of nerve repair, coaptation, grafting, transfer, or decompression, a sterile HPTC collagen membrane is hydrated as per manufacturer instructions, trimmed to the length of the treated nerve segment (approximately 1.5-4 cm), and wrapped circumferentially as a loose perineural sleeve. The wrap is secured using fibrin glue or fine absorbable sutures. Standard wound closure and postoperative rehabilitation protocols are followed.

SUMMARY:
This prospective multicentre observational registry evaluates early clinical outcomes following the use of High-Purity Type I Collagen (HPTC) as a circumferential nerve wrap during peripheral nerve procedures. Eligible procedures include nerve repair, coaptation, grafting, nerve transfers, and decompressions in the upper and lower limbs.

Primary outcomes include early motor recovery assessed using the Medical Research Council (MRC) motor grading system. Secondary outcomes include sensory recovery, neuropathic pain, patient-reported functional outcomes, complication rates, and patient satisfaction assessed at standardized postoperative intervals up to two months.

DETAILED DESCRIPTION:
Peripheral nerve surgery outcomes are often compromised by perineural fibrosis, neuroma formation, and unpredictable axonal regeneration. High-Purity Type I Collagen (HPTC) is a bioengineered resorbable collagen membrane designed to act as a biologic scaffold and perineural barrier, potentially reducing scar adherence and facilitating nerve gliding.

This prospective registry enrolls adult patients undergoing peripheral nerve procedures where HPTC is used as an adjunct circumferential nerve wrap. Functional motor recovery, sensory recovery, pain scores, patient-reported outcomes, and complications will be systematically documented at baseline and follow-up intervals up to four months. This registry aims to generate real-world, multicentre evidence regarding the safety and early clinical effectiveness of HPTC nerve wrapping.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Patients undergoing peripheral nerve procedures including: Primary nerve repair, Nerve coaptation, Nerve grafting, Nerve transfer, Revision nerve decompression
* Upper or lower limb nerve involvement
* Intraoperative use of HPTC nerve wrap
* Ability to comply with follow-up
* Written informed consent provided

Exclusion Criteria:

* Active infection at the surgical site
* Known hypersensitivity to collagen products
* Severe uncontrolled systemic illness
* Pregnancy or lactation
* Re-operation at the same nerve site within the previous 6 months
* Inability to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Motor Functional Recovery | 2 months post-operative
  Motor recovery of the involved muscle groups assessed using the Medical Research Council (MRC) Motor Grading system. Outcome is defined as the proportion of patients achieving MRC grade ≥ M3.
Sensory Recovery - Static and Moving Two-Point Discrimination | 2 months post-operative
  Sensory recovery assessed using static and moving two-point discrimination testing in the affected nerve distribution, measured as the minimum distance (in millimeters) at which two points are perceived as separate.
Sensory Recovery - Semmes-Weinstein Monofilament Sensory Threshold | 2 months post-operative
  Sensory recovery assessed using Semmes-Weinstein monofilament testing in the affected nerve distribution, reported as the lowest monofilament force perceived by the patient.

SECONDARY OUTCOMES:
Neuropathic Pain Intensity | 1 month and 2 months post-operative
  Neuropathic pain intensity measured using the Visual Analog Scale (VAS), where 0 represents no pain and 10 represents worst imaginable pain.
Upper Limb Patient-Reported Functional Outcome (QuickDASH) | 1 month and 2 months post-operative
  Upper limb function assessed using the Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire. The QuickDASH consists of 11 items scored on a scale from 0 to 100, where 0 represents no disability and 100 represents maximum disability. Higher scores indicate worse functional outcome.
Lower Limb Patient-Reported Functional Outcome (LEFS) | 1 month and 2 months post-operative
  Lower limb function assessed using the Lower Extremity Functional Scale (LEFS). The LEFS consists of 20 items with a total score ranging from 0 to 80, where higher scores indicate better functional outcome.
Postoperative Complications | Up to 2 months post-operative
  Incidence of postoperative complications including surgical site infection, neuroma formation, need for re-exploration, or foreign body reaction related to the collagen wrap.
Patient Satisfaction | 2 months post-operative
  Patient satisfaction assessed using a 5-point Likert Satisfaction Scale, with scores ranging from 1 (very dissatisfied) to 5 (very satisfied). Higher scores indicate greater patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Prema Dhanraj, MS, MCh, Study Chair — Rajarajeshwari Medical College and Hospital
Locations (2):
- India (2):
  - Adichunchanagiri Institute of Medical Sciences, Mandya, Karnataka
  - Mysore Medical College and Research Institute, Mysore, Karnataka

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported for the primary and secondary outcomes of this study, including motor recovery scores (MRC grading), sensory assessment results, pain scores (VAS), patient-reported outcome measures (QuickDASH/LEFS), complication data, and relevant baseline demographic and procedural variables.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be made available beginning 6 months after publication of the primary study results and will remain available for up to 5 years following publication.
Access Criteria: Access to the de-identified IPD will be granted to qualified researchers who submit a methodologically sound research proposal. Requests will be reviewed by the principal investigator and study steering committee. Data will be shared under a data-sharing agreement to ensure protection of participant confidentiality.

REFERENCES:
- [Background] Klein S, Vykoukal J, Felthaus O, Dienstknecht T, Prantl L. Collagen Type I Conduits for the Regeneration of Nerve Defects. Materials (Basel). 2016 Mar 23;9(4):219. doi: 10.3390/ma9040219. PMID 28773346
- [Background] Kokkalis ZT, Mavrogenis AF, Ballas EG, Papagelopoulos PJ, Soucacos PN. Collagen nerve wrap for median nerve scarring. Orthopedics. 2015 Feb;38(2):117-21. doi: 10.3928/01477447-20150204-04. PMID 25665110
- [Background] Tanaka H, Kurimoto S, Hirata H. Efficacy of collagen conduit wrapping with collagen fibers on nerve regeneration in sciatic nerve injury with partial transection: An experimental study in the rat model. J Biomed Mater Res B Appl Biomater. 2024 Jan;112(1):e35369. doi: 10.1002/jbm.b.35369. PMID 38247253
- [Background] Narayan N, Shivannaiah C, Gowda S. Evaluating the Efficacy of High-Purity Type I Collagen-Based Skin Substitute Versus Dehydrated Human Amnion/Chorion Membrane in the Treatment of Venous Leg Ulcers: A Randomized Controlled Clinical Trial. Cureus. 2025 Jul 30;17(7):e89031. doi: 10.7759/cureus.89031. eCollection 2025 Jul. PMID 40747200
- [Background] Narayan N, Ramegowda YH, Raghupathi DS, Chethan S, Gowda S. Biological Skin Substitutes in Pressure Ulcers: High-Purity Type I Collagen-Based Versus Amnion/Chorion Membrane. Cureus. 2025 Aug 25;17(8):e90956. doi: 10.7759/cureus.90956. eCollection 2025 Aug. PMID 40862036
- [Background] Narayan N, Shivaiah R, Kumar V, Kumar KM, Chethan S, Gowda S. Comparative Efficacy of High Purity Type I Collagen-Based Skin Substitute and Dehydrated Human Amnion/Chorion Membrane in Diabetic Foot Ulcers: A Multicentre Randomized Controlled Trial. Cureus. 2025 Oct 19;17(10):e94952. doi: 10.7759/cureus.94952. eCollection 2025 Oct. PMID 41122365
- [Background] Narayan N, Raghupathi D, Ramamurthy V, Chethan S, Gowda S. A Comparative Analysis in the Treatment of Full-Thickness Wounds: Negative-Pressure Wound Therapy (NPWT) Combined With High-Purity Type I Collagen-Based Skin Substitute Versus NPWT Alone. Cureus. 2025 Nov 16;17(11):e96977. doi: 10.7759/cureus.96977. eCollection 2025 Nov. PMID 41250786
- [Background] Lee S, Ahmad A, Jeon G. Combining Bootstrap Aggregation with Support Vector Regression for Small Blood Pressure Measurement. J Med Syst. 2018 Feb 28;42(4):63. doi: 10.1007/s10916-018-0913-x. PMID 29488105
- [Background] Mayrhofer-Schmid M, Klemm TT, Aman M, Kneser U, Eberlin KR, Harhaus L, Boecker AH. Shielding the Nerve: A Systematic Review of Nerve Wrapping to Prevent Adhesions in the Rat Sciatic Nerve Model. J Pers Med. 2023 Sep 24;13(10):1431. doi: 10.3390/jpm13101431. PMID 37888042
- [Background] Radecka W, Nogalska W, Siemionow M. Peripheral Nerve Protection Strategies: Recent Advances and Potential Clinical Applications. J Funct Biomater. 2025 Apr 24;16(5):153. doi: 10.3390/jfb16050153. PMID 40422818